CLINICAL TRIAL: NCT06711159
Title: SLEEPINESS - a Search for a Biomarker of Excessive Daytime Sleepiness in Severe Obstructive Sleep Apnoea - An Explorative Study
Status: Recruiting | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: UNEEG Medical A/S (Industry); T&W Engineering A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: EMN-2021-06803
Record Dates: First submitted 2024-11-03; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea (OSA); Excessive Daytime Sleepiness
Keywords: Excessive daytime sleepiness; Ultra long-term EEG; Obstructive Sleep Apnea; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: continuous positive airway pressure — Initiation of treatment with continuous positive airway pressure for obstructive sleep apnea

SUMMARY:
Study aim:

This study aims to use a new brainwave monitoring device that meassure brainwaves 24 hours a day to create better understanding of sleep-wake interplay as a biomarker for excessive daytime sleepiness because of obstructive sleep apnea.

Study Method, Design, and Procedures Patients with sleep apnea referred to the Sleep Clinic at the Department of Ear, Nose, Throat, and Jaw Surgery in Køge for CPAP treatment, who also experience severe daytime sleepiness, will be offered participation in this study. The goal is for 15 participants to complete the entire protocol.

Procedure Overview Initial Sleep Assessment: The study begins with an in-depth sleep assessment through polysomnography (PSG) followed by a Multiple Sleep Latency Test (MSLT).

PSG: This sleep study evaluates sleep structure, confirms sleep apnea, and rules out other sleep disorders.

MSLT: This test measures the brain's tendency to fall asleep during the day. Additional Home-Based Sleep Studies: Participants will undergo two more PSG studies in their homes.

EEG Monitoring: After the initial assessments, participants will have a small EEG electrode implanted to monitor brain activity.

The implant, a CE-certified device called 24/7 EEG™ SubQ, will be inserted under local anesthesia by an experienced surgeon.

Once post-surgery swelling subsides (after about 7-10 days), continuous EEG monitoring will begin, where participants connect an external data storage device during the day. The device records for 12 weeks, and CPAP treatment begins around the 6-week mark.

After 12 weeks, the EEG device is removed, and the study ends. Aditional Data Collection (Optional)

During the 12 weeks of EEG recording, participants are asked to report:

Sleep Diary: Log daytime sleep episodes, including planned naps and unintended naps.

Questionnaires and Tests: Complete daily questionnaires about fatigue symptoms and perform a brief attention and reaction test. These tasks take 3-10 minutes each day and are accessible via smartphone or tablet.

Interviews and Movement Tracking: Participants may also be invited to interviews on how sleepiness affects their daily life and asked to wear a motion-tracking watch to monitor activity.

DETAILED DESCRIPTION:
2.1 Background Sleep quality and quantity is essential for a healthy life. One prominent spoiler of good sleep quality is sleep fragmentation duo to sleep disordered breathing like obstructive sleep apnoea (OSA). A recent global estimation of OSA prevalence estimated that close to 1 billion people suffer from OSA. With a global population of advancing age and increasing obesity the global OSA prevalence seems at a rise.

The health-related consequences of OSA are many; Surge towards metabolic syndrome and an increased cardiovascular risk is well established within the scientific literature. But very invalidating is the inability to obtain restorative sleep through the night and its daytime fellow excessive daytime sleepiness (EDS) which is a key feature for some OSA patient. This reduces quality of life, work ability and general cognitive function as well as driving performance. Furthermore EDS has been is linked to increased comorbidity and mortality.

The American Academy of Sleep Medicine (AASM) defines EDS as "the inability to maintain wakefulness and alertness during the major waking episodes of the day, with sleep occurring unintentionally or at inappropriate times almost daily for at least three months"

3 Study design - overview 3.1 Description of study design This study is an exploratory study in severe OSA patients with EDS defined as an ESS > 10 to record ultra-long-term EEG data with a subcutaneous EEG electrode 6 weeks prior to starting CPAP treatment and 6 weeks after initiation of CPAP treatment. The scope is to detect and quantify episodes of sleep phenomena during normal daytime and study CPAP related sleep rehabilitation.

The hypothesis is that the recordings will show episodes of daytime lapses into sleep both registered by the subject but also episodes of EEG recordings with sleep phenomena that will not be registered by the subject. We hypothesise that CPAP treatment will decrease the quantity of these events in a dose dependant manner. Can this be used as a biomarker for EDS in OSA patients? Is this biomarker stable for patients who do not experience a reduction in ESS when they start CPAP? Will the reduction in EEG recorded sleep phenomenons follow a reduction in other sleepiness scores or sleepiness related cognitive performance? The study period will be running over a period of approximately 4 months from inclusion to completion of the study. The subject enrolled will follow the ordinary patient flow for new referrals within the sleep clinic. The participation in the study will not postpone the timeframe within the OSA patient normally starts CPAP treatment.

Subjects will be recruited after a new referral to the sleep clinic with a diagnosis of OSA and ESS > 10 and screened according to criteria of inclusion and exclusion. Eligible subjects will be enrolled and will start CPAP treatment within the ordinary waiting time to start OSA treatment. Up to 25 subjects are planned to be enrolled to ensure 15 subjects completing the study.

The subjects will start the study by a full PSG test followed by a MSLT. If the result of these test is in conflict with the criteria of inclusion and exclusion the subject will be excluded from the further study.

The subjects will have the UNEEG™ SubQ implanted (the implant) (see "24-7 EEG™ SubQ") and after approximately 10 days of healing, the study subjects will start wearing the 24/7 EEG™ SubQ as much as possible the following 12 weeks. Two secondary PSG will be performed after implantation. The first prior to OSA treatment initiation and the second after treatment initiation.

Sleep diary, subjective sleepiness scores and cognitive test During the study period the subjects will be asked to complete a sleep diary with registration of episodes of daytime napping (intended and unintended).

Subjects will be asked to fill out subjective scores of sleepiness (e.g. Epworth and Karolinska sleepiness scale) on a daily basis during the study period as well as completing a simple cognition test on a tablet or telephone such as a psychomotor vigilance task test (PVT) lasting 3-10 minutes.

Subjects will be invited to participate in scientific semi-structured interviews focusing on the everyday life burden of chronic sleepiness in relation to obstructive sleep apnea and the treatment related rehabilitation from chronic sleepiness.

This study will be conducted in accordance with this investigational plan, ethics committee requirements, the Declaration of Helsinki and applicable local governmental regulations.

5.5 Withdrawal criteria The subject may withdraw at will at any time without explanation. The subjects may be withdrawn from the study at the discretion of the investigator due to a safety concern or if judged non-compliant with the study procedures.

Subjects must be withdrawn from the study for any of the following reasons:

1. Included in the study in violation with any of the inclusion and/or exclusion criteria.
2. The subjects may be withdrawn from the study at the discretion of the investigator due to a safety concern or if judged non-compliant with the study procedures.

Withdrawal will not impact any treatment or follow-up of the subject. Although a subject is not obliged to give his/her reason(s) for withdrawal, the investigator must make a reasonable effort to ascertain the reason(s), while fully respecting the subject's rights.

6 Methods and assessments

This clinical trial will consist of 7 visits from inclusion to completion. The visits are labeled as the following and the specific study activities and visits will be described in details below.

1. Inclusion
2. Pre-PSG and MSLT
3. Implantation
4. Start-up
5. PSG
6. 6 week recording, START CPAP
7. PSG
8. 12 weeks recording and device explantation
9. Follow-up, end of study This clinical trial will take place at Zealand University Hospital Department of Otorhinolaryngology and Maxillofacial Surgery (Køge) Department of Neurology, Roskilde All activities will be under the responsibility of the principal investigator.

   During all study related activities the subjects will be insured by the patient insurance of Zealand University Hospital (Patienterstatningen).

   Patient related information described in the following will be obtained by medical interviewing and will be confirmed for data source identification reasons by a look up in the subject's patient file.

   6.1 Description of study activities and procedures

   6.1.10 EEG recording device for ultra-long-term EEG recordings The ultra-long-term (>2 weeks) EEG recordings will be made using the 24/7 EEG™ SubQ, a CE approved device manufactured by UNEEG™ Medical A/S, Nymøllevej 6, 3540 Lynge, Denmark.

   The electrode will be implanted behind the ear with the electrode positioned over the temporal lobe. The side is chosen at the one that the patient most often do not sleep on. The subjects will be instructed in mounting and using of 24/7 EEG™ SubQ (according to the instruction for use) every night during sleep in the study period. The subjects will asked to create an event by double-tapping the power button on the logger twice when they intentionalley take a nap. The subjects will asked to create an event by double-tapping the power once when the recognice they wake up from an unintended nap.

   The implantation and explanation of the device, postoperative assessment and suture removal will take place at the Department of Otorhinolaryngology and Maxillofacial Surgery (Køge).

   6.1.1 PSG and MSLT The PSG will be mounted by trained personnel on a study site and performed according to the AASM criteria for PSG mock-up. The PSG night recordings will be made in an outpatient setting where the subject sleep in their own home. The day after the subjects will meet on site for the MSLT. The MSLT study protocol will follow the AASM guideline. Thereafter the PSG equipment will be demounted. The PSG/MSLT recordings will be performed with CE approved equipment. The PSG and MSLT data analysis will be conducted by a trained sleep technician according to the AASM criteria and evaluated by a physician with expertise in sleep medicine. The clinically relevant results of the PSG and MSLT will be given to the subject by a medical doctor at the following in-site visit. If the results of the PSG is in violation with the inclusion criteria the subject must be excluded from the study before implantation of the subcutaneous EEG devise.

   6.1.2 Sleep diary The study subjects should fill out the sleep diary every evening prior to going to bed focusing on episodes during the day with all experienced episodes of daytime sleeping or dozing off. The study subjects will be asked to mark every episode as either intentional napping (I) or unintentional napping (U) in the sleep diary.

   6.1.3 Photo of implant area Photos of the area where the implant is located will be taken at visit 3 and 6. The photos will be taken at different angles and distances in combination with one or more fiducial markers. The photos will be taken such that facial recognition is not possible.

   6.1.4 Patient-reported outcome measures and Cognitive test During the study period the study subjects will be asked to perform Patient-reported outcome measures (PROM) evaluating sleepiness symptoms on a daily basis(e.g. 08:00; 11:00, 15:00, 19:00, 22:00). Measures like the Epworth Sleepiness Scale (ESS), a 4-point likert scale where the subject rates the likelihood of them dozing of or falling asleep and the Karolinska Sleepiness Scale (KSS), a 9 point scale raging from 1 "extremely alert" to 9 "very sleepy, great effort to keep alert, fighting sleep" will be used. In relation to the sleepiness PROM the subjects will be asked to perform a simple cognitive test measuring cognition processes like reaction time and alertness. The PROM and the cognitive test takes approximately 5-10 minutes to perform. The data collection for these data will be performed on a tablet or smartphone and supported by a data collection service like www.carp.cachet.dk.

   CARP Cognition Package - Copenhagen Research Platform (CARP) (cachet.dk) Here the relevant cognitive test can also be found called "Reaction Time".

   6.1.5 Actigraphy During the study period the study subjects will be asked to wear an actigraphy unit measuring gross motor activity. The unit will be a wristwatch-like device for monitoring physical rest/activity.

   6.1.6 Interview During the study period the study subjects will be invited to participate in interviews focusing on sleepiness symptoms in relation to everyday life before and after treatment initiation.

   6.2 Other baseline assessments 6.2.1 Demographics

   The following demographics will be recorded at visit 1 and recorded in the case report form CRF:
   * Date of birth
   * Sex
   * Height
   * Weight
   * Profession
   * Preferred sleeping position
   * Preferred sleep duration and time of the day

   6.3 Description of study visits Recruitment and information visit New referrals to the sleep clinic that is fund eligible to the study inclusion criteria (age > 18y, severe OSA and ESS > 10) will be contacted and asked permission to send study information. Patients will be asked to contact the clinic if they find the study interesting and would like to hear more. Interested patient will be invited to an information visit and will be informed about the opportunity to bring a close relative.

   At the individual information visit the information will be given in a simple language and by an undisturbed medical doctor (field-investigator). The oral information will be according to the information given in the "Deltagerinformation_SLEEPINESS" and will take place in a private office. The subjects will be given the opportunity to ask questions regarding the study. Subjects will be given the informed consent form. Subjects will be given a minimum of 3 days reflection time to consider participation. If subjects decide to participate they will sign and hand in the informed consent form and will thereafter be invited to Visit 1: inclusion.

   The subject must sign and date the informed consent form and authority declaration prior to any study related activities.

   Subjects will be screened according to the inclusion and exclusion criteria. 6.3.1 Visit 1: Inclusion This visit can be a telephone visit or in site visit. Check inclusion and exclusion criteria

   • Record concomitant medication, demography, medical history, ESS-score. If the subject is confirmed eligible, the time of implantation should be scheduled.

   6.3.2 Visit 2: Pre-PSG and MSLT This visit will be scheduled to take place around 1 weeks after inclusion.

   The following will be performed and recorded in the CRF:
   * Check withdrawal criteria and record changes in concomitant medication
   * Produce ESS score
   * Perform PSG and following MSLT 6.3.3 Visit 3: Implantation Implantation of the 24/7 EEG™ SubQ will take place at Zealand University Hospital.

   The subject does not need to meet in a fasting condition. The implantation will be performed by a surgical procedure under local anaesthetic.

   The following will be performed and recorded in the CRF:
   * Check withdrawal criteria and record any AEs, or changes in concomitant medication since last visit.
   * Implant UNEEG™ SubQ

   In addition:

   • Dispense information sheet regarding postoperative precautions and give instructions as needed.

   6.3.4 Visit 4: Start-up visit This visit will be scheduled to take place 8-12 days after site visit 3. The site of implantation will be inspected, and sutures removed by trained personnel.

   Dispense external parts of 24/7 EEG™ SubQ including an external data storing unit, adhesive pads and charger. The subject must be instructed in how to mount the device correctly behind the ear, how to use the functionality of the device and how to charge the battery according to the patient instruction for use (also dispensed). Find a suitable time for a 24 hour PSG within the following 6 weeks.

   The following will be performed and recorded in the CRF:

   • Check withdrawal criteria and record any AEs and any changes in concomitant medication since last visit.
   * Dispense sleep diary and give instructions
   * Dispense 24/7 EEG™ SubQ and give instructions
   * Dispense videorecorder and give instructions
   * Produce ESS and KSS score and PVT

   In addition:

   Take close-up photos of the area where the implant is located 6.3.5 Visit 5: PSG This visit will be scheduled to take place between week 1-6 after visit 4.

   The following will be performed and recorded in the CRF:

   • Check withdrawal criteria and record changes in concomitant medication
   * Produce ESS score and KSS score and PVT
   * Perform ambulant 24 hours PSG 6.3.6 Visit 6: 6 week recorded, Start CPAP This visit will be scheduled to take place at the study site 6 weeks after visit 4.

   The following will be performed and recorded in the CRF:
   * Download data from 24/7 EEG™ SubQ
   * Check withdrawal criteria and record any AEs and any changes in concomitant medication since last visit.
   * Record any device deficiencies since last visit

   In addition:

   • Collect and review sleep attack diary

   • Produce ESS and KSS score and PVT.

   Subjects will be educated in the use of CPAP by a trained personnel according to the standard of handing out CPAP within the sleep clinic. Dispense of CPAP machine and mask.

   6.3.7 Visit 7: PSG This visit will be scheduled to take place between week 1-6 after visit 6.

   The following will be performed and recorded in the CRF:

   • Check withdrawal criteria and record changes in concomitant medication
   * Produce ESS score and KSS score and PVT
   * Perform ambulant 24 hours PSG

   6.3.8 Visit 8: 12 week recording, device explantation, end of study. This visit will be scheduled to take place 6 weeks after visit 4.

   The following will be performed and recorded in the CRF:

   • Download data from 24/7 EEG™ SubQ
   * Check withdrawal criteria and record any AEs and any changes in concomitant medication since last visit.
   * Record any device deficiencies since last visit

   In addition:
   * Collect and review sleep attack diary
   * Produce ESS and KSS score and PVT
   * Explant 24/7 EEG™ SubQ The subject does not need to meet in a fasting condition. The explantation will be performed by a surgical procedure under local anaesthetic. More information is available in the instruction for use.

   6.3.9 Visit 9: Follow-up This visit will be scheduled to take place 7-10 days after visit 6. The site of explanation will be inspected, and sutures removed by trained personnel. Any AEs or changes in concomitant medication since last visit will be recorded in the CRF. Produce ESS and KSS score and PVT.

7 Study safety 7.1 Adverse events and adverse device effects At all study visits any adverse event (AE) and adverse device effect (ADE) as well as serious adverse event (SAE) and serious adverse device effect (SADE) will be evaluated by sub-investigator (MD and PhD running the study), reported in the CRF, assessed of intensity and expectedness, clinically cared for and followed up until the outcome of the event is "recovered", "recovered with sequelae" or "fatal", and until all queries have been resolved.

7.2 Early termination or suspension of the investigation If the investigator finds continuation of the study incompatible with the safety of the study subjects due to any safety related issues of the study device or the study procedure, the study will be terminated or postponed until these issues have been solved.

If a study is prematurely terminated or suspended, the investigator should promptly inform the subjects and assure appropriate follow-up. Furthermore, the investigator should promptly inform the ethics committee and provide a detailed written explanation. The regulatory authorities should be informed according to the regulations.

8 Statistical considerations and data reporting As this is an exploratory and observational study per design a similar exploratory approach will be used when it comes to statistical analysis. Therefore the statistical analysis plan is not fixed and the choice of statistical methods will be data dependant. Power analysis is not possible given the circumstances.

Data will be scrutinized for potential biomarkers related to EDS. The data analysis will be conducted in collaboration with the Technical University of Denmark (DTU). The preliminary approach is based on classical time domain and frequency domain analysis. The use of artificial intelligence (AI) and/or machine learning (ML) will be used when applicable.

8.1 Rational for the choice of sample size Previous studies in sleepiness quantification have shown considerable intra-individual variability. (14) When taken this in account when choosing sample size, 15 subjects completed seem a fair number to collect enough data to be able to evaluate the use of subcutaneous EEG recordings for OSA patients with EDS as well as not too little to get a representative sample size. To obtain 15 successful datasets we expect to include up to 25 individuals due to expected failures of a diversity of reasons.

9 Ethics The study will be conducted according to the declaration of Helsinki, and approved by the local ethics committee. Only information relevant for the study will be collected. Data will be handled in accordance with the General Data Protection Regulation and Data Protection Act as well as Danish data protection law.

9.1 Subject benefit and risks All medical device equipment used for this study protocol will be used in accordance with the instruction for use and contraindications for the medical devices have been included in the exclusion criteria.

Subjects within this study will get the opportunity to get an in depth evaluation of their sleep quality as well as an objective test for sleepiness (PSG and MSLT). These test are resource intensive and because of that few OSA patient get the opportunity to be evaluated by such test.

The following side effects for 24/7 EEG™ SubQ are listed in the instruction for use:

"General side effects normally associated with any surgical implantation procedure or local anesthesia also apply to the placement of the implant.

Specifically, you may experience the following side effects with the implantation and use of the system:

* Up to 3 weeks after the surgical procedure, hematoma or seroma may appear near the implant.
* Temporary pain, headache, infection and discomfort (including soreness, inflammation, swelling, irritation and itching) may appear around the implant up to 3 weeks after the surgical procedure.
* Wound healing may be compromised.
* Infection, swelling, soreness, irritation or itching of the skin around the implant.
* Occasional headache or pain during long-term use of the system."

No radioactive substances are used in the study. 9.2 Ethical considerations Since obstructive sleep apnoea increases the risk of motor vehicle accidents and sleepiness related accidents are potentially preventable it is important to continually evaluate the OSA patient for fitness to drive. (6) This is a difficult evaluation and clinicians have few unreliable objective measures to guide this evaluation. As this study will shed light on wake/sleep transition in OSA patients everyday life it might provide us with better knowledge on how to determine fitness to drive and therefor possible enhance road safety in the future.

The implantation of the 24/7 EEG™ SubQ device is seen as a minor surgical procedure with a limited risk of complications and side effects. It is estimated that the overall aim of this study outweighs the burden the study inevitably will put on the study subjects.

9.3 Changes to clinical investigation plan or related procedures Major design changes in the clinical investigation including amendment to the clinical investigation plan, informed consent, or other written information provided to subjects, and/or study procedures directly must be approved in writing by the ethics committee before implementation.

9.4 Deviations from clinical investigation plan Deviation to the clinical investigation plan should be avoided. Significant deviations compromising or potentially compromising the safety of the subjects, enrolment of non-eligible subjects or any deviation, which significantly compromises the outcome of the study, must be reported to the ethics committee within the appropriate timelines indicated by the ethics committee.

9.5 Reporting of results The findings of the study will be published in international peer reviewed journals. Furthermore, they (positive, negative or inconclusive) will be made publicly available in the European Database on Medical Devices (EudaMed) or the North American www.clinicaltrials.gov.

First author will be Mathias Sarkez-Knudsen and last author will be and Preben Homøe alternating Martin Ballegaard according to the primary context.

9.6 Conflict of interest and financial support The study is initiated by the primary investigator Professor Preben Homøe, and sub-investigator Mathias Sarkez-Knudsen from the department of Otorhinolaryngology in collaboration with associate professor Martin Ballegaard from the department of neurology.

UNEEG medical a/s and T&W a/s has been invited to participate in the project and will deliver device knowledge and data science qualifications to support the data analysis.

The study is financed by the EU INTERREG ØKS (Øresund, Kattegat og Skagerak) as part of the project InnoSleep. InnoSleep is financing the salary of the Ph.D. student (aprox. 240.000€) and the study equipment (aprox. 210.000€) as well as the other study expenses (aprox. 59.000€).

None of the investigators report any conflict of interests.

ELIGIBILITY:
Inclusion Criteria:

For a subject to be eligible, all inclusion criteria must be answered "yes":

1. Age ≥18 years
2. Subjects must be diagnosed with Severe Obstructive Sleep Apnea (AHI > 30) and have not yet started any form of PAP (positive airway pressure) treatment.
3. ESS score must be above 10 at the time of inclusion.

Exclusion Criteria:

For a subject to be eligible, all exclusion criteria must be answered "no":

1. Known severe neurological or psychiatric diseases.
2. Known congestive heart failure, chronic renal failure, liver failure, malignancy, severe pulmonary disease.
3. Considerable use of alcohol.
4. Medication judged by investigator to influence sleep/wake regulation to such a degree that data quality will be compromised.
5. Has cochlear implants.
6. Involved in therapies with medical devices that deliver electrical energy into the area around the implant.
7. Is at high risk of surgical complications, such as active systemic infection and haemorrhagic disease.
8. Are unable (i.e. mentally or physically impaired patient), or do not have the necessary assistance, to properly operate the device system.
9. Has an infection at the site of device implantation.
10. Operates MRI scanners.
11. Has a profession/hobby that includes activity imposing extreme pressure variations (e.g. diving or parachute jumping). NB: diving/snorkelling is allowed to 5 metres depth.
12. Has a profession/hobby that includes activity imposing an unacceptable risk for trauma against the device or the site of implantation (e.g. martial art or boxing).
13. Other known diseases or conditions, judged by investigator to influence sleep to such a degree that data quality will be compromised.
14. Incapable, judged by the investigator, of understanding the participant instruction or who are not capable of carrying through the investigation.
15. Pregnancy or intention to become pregnant within the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for this study are patients who suffer from Excessive Daytime Sleepiness (defined by an epworth sleepiness scale above 10 at inclussion) because of untreated Obstructive Sleep Apnoea (OSA) and with the inclusion/exclusion criteria listed below to ensure generalizability of study and to minimize the influence of other contributors to EDS.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-10-11 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultra long-term EEG derived sleepiness biomarker | From enrollment to completion 4 months
  Our primary explorative objective is to scrutinize subcutaneous Ultra Long-term EEG for potential biomarkers predicting sleepiness in OSA patients. Determining daytime wake-to-sleep transition rate, episodes of microsleep, and episodes of macro sleep, alongside the duration and patterns of these events. Our explorative findings will be correlated and preliminary validated against the well-established sleepiness metrics and questionnaires, multiple sleep latency test (MSLT), Epworth Sleepiness scale (ESS), Karolinska Sleepiness Scale (KSS), and a 3-minute psycomotor vigilance tast test (PVT), as well as to the patient's experience of falling asleep or dozing off intentionally and unintentionally in the form of a "sleep and nap diary". Any potential sleepiness biomarker derived from this study will be available for future confirmatory trials.
The effects of CPAP treatment on ultra long-term EEG | From enrollment to completion 4 months
  Our experimental objective is to determine the effects of CPAP treatment on sleep quality, quantity, and timing from the day-to-day perspective that ULT-EEG provides. Furthermore, the experimental design enables us to clinically validate the exploratively deduced sleepiness biomarker candidates through comparisons before and after the intervention of CPAP treatment conditions. Previous studies on the effect of CPAP on sleepiness reduction have shown a dose-dependent configuration with CPAP usage. ESS is typically reduced by 4,78 (or more). We expect relevant biomarker candidates to follow similar patterns when CPAP is introduced in a population with severe OSA and EDS.

SECONDARY OUTCOMES:
Validate automatic sleep/wake classification from ultra long-term EEG for patients with severe obstructive sleep apnea | From enrollment to completion 4 months
  Our Secondary objective is to validate automatic sleep/wake classification based on two-channel subcutaneous EEG against golden standard manually scored polysomnography in patients with severe OSA. Additionally, we explore the use of Ecological Momentary Assessment (EMA) methods to record Excessive Daytime Sleepiness in OSA.

CONTACTS AND LOCATIONS:
Overall Officials: Preben Homøe, Professor, Principal Investigator — Zealand University Hospital, Department of Otorhinolaryngology
Locations (1):
- Zealand University Hospital, Koege, Regional Zealand, Denmark

IPD SHARING:
Plan to Share IPD: Undecided